CLINICAL TRIAL: NCT05168722
Title: COVID-19, Patients' Evolution and the Influence of the Pandemic on Health Care and Outcomes in Chronic
Brief Title: COVID-19, Patients' Evolution and the Influence of the Pandemic on Health Care and Outcomes in Chronic Diseases
Status: Completed | Type: Observational
Sponsor: Hospital Galdakao-Usansolo (Other Government)
Collaborators: Instituto de Salud Carlos III (Other Government); European Regional Development Fund (Other)
Responsible Party: Principal Investigator, JOSE M QUINTANA-LOPEZ, MD PhD, Head of the Research Unit, Hospital Galdakao-Usansolo
Other Study IDs: PI21/00824
Record Dates: First submitted 2021-12-22; First posted 2021-12-23 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: COVID-19 Pandemic; Pulmonary Disease, Chronic Obstructive; Heart Failure, Congestive; Depressive Symptoms
MeSH Terms: conditions — COVID-19; Pulmonary Disease, Chronic Obstructive; Heart Failure; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No interventions — No interventions

SUMMARY:
Objectives: 1.- To evaluate the changes in health care and use of services in patients with chronic diseases such as chronic obstructive pulmonary disease (COPD), heart failure and major depression between 2017-2019 and the years 2020-2022, COVID pandemic period, and to see their relationship with clinical outcomes (in terms of mortality, admissions, death, current situation of his disease) and changes in health-related quality of life. 2- To evaluate the health care provided to a cohort of patients diagnosed with SARSCOV-2 (COVID-19 positive) during 2020 based on accessibility, equity and outcomes obtained. 3-To evaluate the evolution of the cohort of patients diagnosed with SARSCOV-2 after two years of follow-up since their diagnosis and create clinical prediction rules for the persistence of symptoms.

Methodology. Four cohorts already created in previous projects are included: three of chronic patients, COPD, heart failure, major depression, all of 2017, and for which baseline information is available for follow-up of the health care they received in the 2017-19 period compared to that received during the 2020-22 period and to see the changes in their health-related quality of life from baseline based on generic and specific questionnaires for each of the pathologies included. Another cohort of positive and admitted patients for COVID-19 in 2020 is included, in whom the services received will be evaluated and recorded symptoms persistency that may have had up to two years after their index admission to develop tools for predicting the persistence of symptoms in the medium-long term.

DETAILED DESCRIPTION:
DESIGN. Cohort study with prospective follow-up of 4 preformed cohorts between years 2017 and 2020 which will be followed until 2022.

SUBJECTS OF STUDY. SELECTION CRITERIA. DESCRIPTION OF THE COHORTS OF CHRONIC PATIENTS.

1. - COHORT OF PATIENTS WITH HEART FAILURE (HF) (Clinicaltrials.gov # NCT03300791).

   Selection criteria: A. Inclusion criteria: patients admitted for insufficiency syndrome acute cardiac arrest including acute (de novo) heart failure and heart failure (HF) previously diagnosed but that has a progressive or rapid worsening of symptoms that requires urgent intervention. (ICD-9 code: 428.x; some of 402.x). Patients over 18 years. Patients who agree to participate and sign the informed consent.

   B. Exclusion criteria: a) patients who develop an episode of HF during admission, if they have been admitted for another reason, b) patients transferred from other health centers c) myocardial infarction or cerebrovascular accident in the 4 weeks prior to admission, d) life expectancy less than one year, due to HF in terminal state or due to a different cause according to the assessment of the study physicians e) impossibility to complete the questionnaires or with external help (reviewer, family, social help) due to sensorineural cause, dementia or lack of knowledge of the language

   Scope: Participating hospitals: Basurto (Bilbao), Donostia (San Sebastian), and Galdakao-Usansolo (Galdakao, Vizcaya). There were 1093 patients. Comité de Ética de la Investigación con medicamentos/ Ethics Committee for Drug Research (CEIm) approval Basque Country baseline study reference PI2015151:
2. - COHORT OF PATIENTS WITH COPD (Clinicaltrials.gov # NCT03227211).

   - Inclusion criteria: episodes of patients with COPD exacerbation who can be admitted with 2 presentations: A) Known case of COPD: Episodes of patients with a previous diagnosis of COPD (FEV1 / forced vital capacity (FVC) <70%) presenting with an exacerbation of COPD. B) New case of COPD: Episodes of patients whose clinical history and anamnesis suspect a COPD: (smokers or ex-smokers of more than 15 packs / year, with basal dyspnea, cough, expectoration for more than three months of the year), who present symptoms compatible with an exacerbation. The diagnosis was confirmed in the pulmonology control consultation within two months after hospital discharge or emergency room, by performing spirometry and always bearing in mind that the patient had to be stable.

   Exclusion criteria: Patients admitted with ventilatory failure obstructive or restrictive due to a different disease (asthma, tuberculosis sequelae, pachypleuritis, restrictive diseases). All COPD cases finally admitted for any other cause, other than exacerbation or complicated COPD. Patients with serious organic or psychopathological problems or in a terminal or neurosensory situation that prevent them from giving their consent and / or completing the questionnaires used in the study. Patients who do not understand the Spanish language and cannot complete the questionnaires. Or that they do not wish to participate or that they do not sign the informed consent that all patients will be passed. There were 1,400 patients from the hospitals of Araba, Donostia, Cruces, Basurto, Santa Marina and Galdakao. CEIm approval Basque Country baseline study reference: 912015124
3. -COHORT OF PATIENTS WITH MAJOR DEPRESSION (ISCIII Reference: PI13 / 00560). Selection criteria. Patients with a diagnosis of depressive disorder (DSM-IV criteria).

Inclusion criteria : patients over 18 years of age diagnosed with depressive disorder, and who after being informed of the objective of the study agree to participate. Exclusion criteria: patients with organic or psychiatric pathologies that prevent them to collaborate in the study; illiterate or patients with sensory deficit that prevent the completion of the outcome measurement instruments included in the study, or patients with bipolar disorder, dysthymia or postpartum depression. There were 433 patients recruited from: Basurto Hospital, Galdakao Hospital, and Mental Health Centers of Basauri, Galdakao, Derio, Uribe, and Ortuella. CEIm approval Basque Country baseline study reference: 12014050) 1.-COHORT OF COVID-19 POSITIVE PATIENTS (Clinicaltrials.gov # NCT04463706). Admitted patients (confirmed cases) of COVID-19 during 2020, excluding the pediatric population. A case of infection by severe acute respiratory syndrome by Corona Virus-2 (SARS-CoV-2) is defined as the one that meets the laboratory criteria: polymerase chain reaction amplification (PCR) positive at a specific gene [RNA-dependent RNA polymerase (RdRp) or S gene] or PCR positive for at least 2 genes used as screening [E or N gene].

SCOPE: Patients admitted for COVID-19 in hospitals in the Basque Country, from 03/01/2020 to on 31/12/2020. There were 3038 patients, 1865 and 1173 registered patients from the first and second wave of the pandemic, respectively. CEIm Basque Country approval baseline study reference: PI2020059.

SAMPLE SIZE. It is based on the previously created cohorts, with sample sizes that range from slightly more than 400 people in the cohort with the smallest sample size to more than 3,000 in the the one that more patients are included.

CALCULATION OF SAMPLE SIZE. Due to the sample sizes that the investigators have in all the cohorts the investigators guarantee being able to respond to the hypotheses of the study with a power of 80% and an alpha error of 0.05 for paired data. Thus, for example, for a decrease in the quality of life of the EuroQol-5D (EQ-5D) of 0.1 points (with a standard deviation of 0.4) 128 people would be needed. Likewise, assuming a change in the proportion of visits that drops by 15% or more would require 165 people for each cohort. In all cases, this estimated sample size is exceeded by our samples. In the case of models predictive predictors of persistence of symptoms, if there is at least 10% of the sample with this persistence of symptoms, with the more than 3000 people in this cohort, this is enough to develop and validate a predictive model.

METHODOLOGY Variables for which the investigators already have information at baseline: In all cases there are sociodemographic data, clinical information (background, associated diseases, level of severity of study disease, baseline treatments, imaging tests, and analytical data when appropriate) and quality of life questionnaires, both generic and specific.

Follow-up. Variables common to all the cohorts that the investigators will collect from the period 2017 to 2019. Apart from the previous baseline information that is already available for each cohort, the investigators will complement it with data on associated diseases to present to patients during this period as well as all prescribed long-term treatments.

Health services use during the study period will be collected on the number of consultations with their primary care physician, primary care nurse, consultations with specialists, participation in telemedicine programs, continuity of care, admission in residence, telematic consultations, laboratory and imaging tests requested, consultations with others specialists, visits to hospital and out-of-hospital emergencies, hospital admissions (with diagnosis at discharge), ICU admissions, or death.

Variables that the investigators will collect in the follow-up until 2022 (including 2020 and 2021) Similarly, the data on the clinical situation of the patients of the various cohorts will be updated.

Information will be collected on the use of social health services during the study period on the number of consultations with their primary care doctor, primary care nurse, consultations with specialists, participation in telemedicine programs, continuity of care, telematic consultations, laboratory and imaging tests requested, consultations with other specialists, visits to hospital and out-of-hospital emergencies, hospital admissions ((with diagnosis at discharge), admissions in ICU, admission to residence, or death.

Variables to be collected in the follow-up of patients diagnosed as COVID positive during the 2020-2022 period. Symptoms that persist over time: fatigue, shortness of breath, cough, joint pain, chest pain, muscle pain or headache, fast heartbeat

, loss of smell or taste, memory problems, concentration or trouble sleeping (insomnia), dizziness tingling, tinnitus, earaches discomfort, diarrhea, stomach pain, loss of appetite, fever, sore throat, rash or hair loss. More serious complications: Cardiovascular: inflammation of the heart muscle. Respiratory: abnormalities in lung function. Renal: Acute kidney injury Dermatological: skin rash, hair loss. Neurological: smell problems and taste, sleep problems, difficulty concentrating, memory problems Psychiatric: depression, anxiety, mood swings. Follow-up tests performed. Imaging tests; function tests pulmonary; of cardiac function. Blood test. Specific treatments established by complications of COVID. COVID vaccination. Time off work (date of incorporation to the job); Need for help (family or social) or admission to a residence.

DATA COLLECTION. All alive patients who agree to participate in this new phase will be contacted. Once they accept and sign the Informed consent, the following sources of information will be used.

* Computer records of tabulated information (data exploitation system in the case of variables which are tabulated: Oracle Analytics Server (OAS)).
* Clinical electronic records: for information that is not indexed in the previous data bases and requires a manual review of the history.

Data mining in OAS will be done by a data analyst. Manual data extraction will perform a data manager, both to be hired in charge of this project, under the supervision of the principal investigator (PI) and clinical collaborators. All data collected by the various sources of information will be entered in a database created in a ad hoc data base, hosted on our administration servers to guarantee their security and confidentiality. Once the information has been extracted from both sources of information, the data analyst will create a common database for further analysis.

STATISTIC ANALYSIS. A descriptive analysis of the entire sample will be carried out (means and standard deviations for continuous variables or frequencies and percentages, for categorical variables) and the differences between the samples of the two times of each cohort will be evaluated by means of the analysis paired data using the paired t or the Wilcoxon paired nonparametric test, if normality is not fulfilled, for continuous variables, and by means of the McNemar test for categorical variables. A univariable analysis will be performed to determine potential factors or variables. related to the outcome variables of interest. Regression will be used for the multivariable analysis conditional logistics or generalized linear models for paired data (GEE). In the case of analysis of unpaired data, the usual statistics for continuous data (t-test, ANOVA) or categorical (Chi-Square, Fisher's exact test). For predictive models, in the case of variables dichotomous dependent (persistent symptoms) multilevel logistic regression models will be used, whose predictive capacity will be measured by the area under the receiver operating characteristic (ROC) curve (AUC) and the calibration of the model using the Hosmer and Lemeshow test; for continuous dependent variables (changes in their quality of life) multilevel generalized linear models will be used. Adjustment variables: diagnostic, severity of the disease, associated diseases, procedures and treatments performed, quality of life related to baseline health. Statistical significance will be assumed when p <0.05 and all Analysis will be carried out using the statistical programs Statistical Analysis System (SAS) v9.4 and R.

ELIGIBILITY:
Inclusion Criteria: patients over 18 years of age diagnosed with depressive disorder, admitted by heart failure or COPD, or positive to COVID-19

-

Exclusion Criteria:

* patients with pathologies organic or psychiatric that prevent collaboration in the study; illiterate or deficit patients sensory that prevent the completion of the outcome measurement instruments included in the study, or who refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Four cohorts already created in previous projects are included, three of chronic patients: 1-COPD, heart failure, major depression , all of 2017, and for which baseline information is available for follow-up of the health care they received in the 2017-19 period compared to that received during the 2020-22 Another cohort of positive and admitted patients for COVID-19 in 2020 is included
Sampling Method: Non-Probability Sample
Enrollment: 2220 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Death | 2 years
  Death during follow up
Health services use | 2 years
  Visits to primary care physician, specialist, outpatient care, emercengy room, hospital admissions
Patient reported outcome measurements changes | 2 years
  Changes in generic and specific patient-reported outcome measure (PROMs) in the study period

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Quintana, PhD, Principal Investigator — Hospital Galdakao-Usansolo
Locations (5):
- Spain (5):
  - Hospital Universitario Araba, Vitoria-Gasteiz, Alava
  - Hospital Galdakao-Usansolo, Galdakao, BIZKAIA
  - Hospital U. Cruces, Barakaldo
  - Hospital U. Basurto, Bilbao
  - Hospital Universitario Donostia, Donostia / San Sebastian